CLINICAL TRIAL: NCT01533272
Title: Open Randomized Study Comparing Two Alternatives of Antiretroviral Therapy as Post-exposure Prophylaxis to HIV-1: TENOFOVIR+EMTRICITABINA + LOPINAVIR/RITONAVIR VS TENOFOVIR+EMTRICITABINA + MARAVIROC
Brief Title: Study Comparing Two Alternatives of Antiretroviral Therapy as Post-exposure Prophylaxis to HIV-1:FOVIR+EMTRICITABINA + LOPINAVIR/RITONAVIR VS TENOFOVIR+EMTRICITABINA + MARAVIROC (MARAVI-PEP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Felipe Garcia, PhD, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MARAVI-PEP
Record Dates: First submitted 2012-02-08; First posted 2012-02-15 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: HIV Infection
Keywords: HIV infection; Postexposure prophylaxis
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; Emtricitabine; Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tenofovir, emtricitabine, Maraviroc (Experimental): New postexposure prophylaxis (it is a combination drug)
  Interventions: Drug: Tenofovir, emtricitabine, maraviroc
- Tenofovir, emtricitabine, lopinavir/r (Active Comparator): Standard prophylaxis (it is a combination drug)
  Interventions: Drug: Tenofovir, emtricitabine, lopinavir/r

INTERVENTIONS:
Drug: Tenofovir, emtricitabine, maraviroc — experimental drug
  Arms: Tenofovir, emtricitabine, Maraviroc
Drug: Tenofovir, emtricitabine, lopinavir/r — Lopinavir/r 400mg BID
  Arms: Tenofovir, emtricitabine, lopinavir/r

SUMMARY:
As a measure of secondary prophylaxis, and with the final objective of avoiding the infection, it has been suggested to use antiretroviral therapy. This is known as post-exposure prophylaxis (PEP).

Although there are different recommendations, almost every guideline recommend using 3 drugs as PEP both in USA and Europe.

Toxicity is one of the main limitations of PEP. Side effects during PEP are very usual, are attributed mainly to PI and are the main reasons for poor adherence or lost of follow-up.

A current standard regimen is AZT+3TC (Combivir®) or tenofovir+emtricitabine (Truvada®) plus the PI lopinavir/r. Toxicity associated with this regimens are high (31-85% of cases), with a 10-35% interruption of PEP Maraviroc, a CCR5 receptor antagonist, very well tolerated, coul be an adequate drug for PEP.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Older than 18 years old
* A potentially sexual exposition to HIV
* Accept to participate

Exclusion Criteria:

* Pregnant women
* The source case a person with HIV antiretroviral resistances
* Persons with a treatment that is contraindicated with the drugs in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2012-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients reaching 28 days of postexposure prophylaxis. | 28 days
  Postexposure prophylaxis has to be used during 28 days to have effectiveness. It is thought that a shorter period of treatment does not prevent HIV infection according to animal models. Therefore, we will assess the proportion of patients who complete the total period of treatment in each arm of the study. The hypothesis is that a higher proportion of patients who take the medication with lower side effects will complete the 28 days of postexposure prophylaxis

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Garcia, PhD, Principal Investigator — Consultant
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Leal L, Leon A, Torres B, Inciarte A, Lucero C, Mallolas J, Laguno M, Martinez-Rebollar M, Gonzalez-Cordon A, Manzardo C, Rojas J, Pich J, Arnaiz JA, Gatell JM, Garcia F; MARAVIPEP Study Group. A randomized clinical trial comparing ritonavir-boosted lopinavir versus maraviroc each with tenofovir plus emtricitabine for post-exposure prophylaxis for HIV infection. J Antimicrob Chemother. 2016 Jul;71(7):1982-6. doi: 10.1093/jac/dkw048. Epub 2016 Mar 18. PMID 26994091